CLINICAL TRIAL: NCT03342443
Title: Effect of Memantine on Radiotherapy-related Cognitive Impairment
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yamei Tang, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20161208
Record Dates: First submitted 2017-05-05; First posted 2017-11-17 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Cognitive Impairment
Keywords: memantine; radiotherapy-related cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- memantine (Experimental): Patients receive memantine with a dosage of 5 microgram at 8 am daily for one week (Week 1), then 5 microgram at 8 am and 5 microgram at 5 pm for one week (Week 2), then 10 microgram at 8 am and 5 microgram at 5 pm for one week (Week 3), then 10 microgram at 8 am and 10 microgram at 5 pm for 21 weeks (Week 4-24), in the absence of unacceptable toxicity or severe deterioration.
  Interventions: Drug: Memantine
- placebo (Placebo Comparator): Patients receive placebo with a dosage of one halfpill at 8 am daily for one week (Week 1), then one halfpillat 8 am andone half pill at 5 pm for one week (Week 2), then one pillat 8 am and one half pill at 5 pm for one week (Week 3), then one pill at 8 am and one pill at 5 pm for 21 weeks (Week 4-24), in the absence of unacceptable toxicity or severe deterioration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Memantine — Patients receive memantine with a dosage of 5 microgram at 8 am daily for one week (Week 1), then 5 microgram at 8 am and 5 microgram at 5 pm for one week (Week 2), then 10 microgram at 8 am and 5 microgram at 5 pm for one week (Week 3), then 10 microgram at 8 am and 10 microgram at 5 pm for 21 weeks (Week 4-24), in the absence of unacceptable toxicity or severe deterioration.
  Other Names: Arm I
  Arms: memantine
Drug: Placebo — Patients receive placebo with a dosage of one halfpill at 8 am daily for one week (Week 1), then one halfpillat 8 am andone half pill at 5 pm for one week (Week 2), then one pillat 8 am and one half pill at 5 pm for one week (Week 3), then one pill at 8 am and one pill at 5 pm for 21 weeks (Week 4-24), in the absence of unacceptable toxicity or severe deterioration.
  Other Names: Arm II
  Arms: placebo

SUMMARY:
Purpose: This randomized, double-blind, placebo-controlled clinical trial aims to evaluate the therapeutic effects of thalidomide in radiotherapy-related cognitive impairment.

Further study details as provided by Sun Yat-sen Memorial Hospital, Sun Yat-sen University / Yameitang.

Primary outcome measure: cognitive improvement, which is determined by the difference value of ADAS-cog score before and after the treatment of memantine.

DETAILED DESCRIPTION:
Application of radiotherapy to patients with head and neck cancer isa mainstay treatment in contemporaryoncology practice. However, patients who received radiation are vulnerable to development of cognitive impairment.There is no acknowledged and effective standard treatment for radiotherapy-related cognitive impairment. We supposed that memantine, as the N-methyl-D-aspartate receptor antagonist, would relieve radiotherapy-related cognitive impairment after head and neck cancer, and would improve the life quality for these patients and their families.

Primary objectives: This randomized, double-blind, placebo-controlled clinical trial aims to evaluate the efficacy of memantineon cognition in radiotherapy-related cognitive impairment.

Secondary objectives:

To evaluate the effect of memantine on sleep disorder, mood disorder, activities of daily living, and safety in patients with radiotherapy-related cognitive impairment.

OUTLINE: This is randomized, double-blind, placebo-controlled clinical trial. Patients will be enrolled and administrated with memantine or placebo. Memantine will be supplied as 10 mg per pill to be taken by mouth. Placebo will be supplied as substitute of 10 mg memantine per pill to be taken by mouth.

Patients will be screened, consented, enrolled and have a washout period for 6 weeks. Then these patients will be randomized to two arms.

Arm І: Patients receive memantine with a dosage of 5 microgram at 8 am daily for one week (Week 1), then 5 microgram at 8 am and5 microgram at 5 pm for one week (Week 2), then 10 microgram at 8 am and 5 microgram at 5 pm for one week (Week 3), then 10 microgram at 8 am and 10 microgram at 5 pm for 21 weeks (Week 4-24), in the absence of unacceptable toxicity or severe deterioration.

Arm ІI: Patients receive placebo with a dosage of one half pill at 8 am daily for one week (Week 1), then one half pill at 8 am and one half pill at 5 pm for one week (Week 2), then one pill at 8 am and one half pill at 5 pm for one week (Week 3), then one pill at 8 am and one pill at 5 pm for 21 weeks (Week 4-24), in the absence of unacceptable toxicity or severe deterioration.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have received radiation therapy due to head and neck cancer.
* Prior irradiation is ≥1.5 yearsand≤ 6 years.
* Age>/= 35 years but age</=60.
* Estimated life expectancy must be greater than 12 months.
* Cognitive impairment exists for more than 4 weeks, withMMSE≤26, or MoCA≤25.
* Routine laboratory studies with bilirubin </=1.0 * upper limits of normal (ULN), aspartate aminotransferase (AST or SGOT) or alanine aminotransferase (ALT)< 1.0 * ULN, creatinine<1.0 * ULN, white-cell count >/= 4,000 per cubic millimeter; neutrophils count >/=1500 per cubic millimeter, platelets >/= 100,000 per cubic millimeter; Hb>/=110 gram per millilitres. PT, APTT, INR in a normal range.
* Constant caregivers who well understand and have willingness to sign a written informed consent document.

Exclusion Criteria:

* evidence of tumor metastasis, recurrence, or invasion;
* evidence of very high intracranial pressure that suggests brain hernia and need surgery;
* previous treatment with memantine or other medications for cognitive impairment;
* history of mental disordersor cognitive impairment before radiotherapy;
* history of stroke, or high risk of vascular dementia;
* family history ofalzheimer's disease, pick's disease, etc.;
* history of severe head trauma;
* clinically significant active disease, e.g. New York Heart Association Grade II or greater congestive heart failure, serious and inadequately controlled cardiac arrhythmia, significant vascular disease, severe infection;
* history of allergy to relevant drugs;
* pregnancy, lactation, or fertility program in the following 12 months;
* participation in other experimental studies.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2017-12-06 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
cognitive improvement | Baseline to Week 24
  Cognitive improvement is determined by the difference value of ADAS-cog score before and after the treatment of memantine.

SECONDARY OUTCOMES:
improvement of global condition | Baseline to Week 24
  Improvement of global condition is determined by the difference values of CIBIC-plus before and after the treatment of memantine.
improvement of activities of daily living | Baseline to Week 24
  Improvement of activities of daily living is determined by the difference values of ADL before and after the treatment of memantine.
improvement of activities of daily living | Baseline to Week 24
  Improvement of activities of daily living is determined by the difference values of Clinical Dementia Rating before and after the treatment of memantine.
improvement of mental statement | Baseline to Week 24
  Improvement of mental statement is determined by the difference values of MMSE before and after the treatment of memantine.
improvement of psychological statement, including sleep disorder, mood disorder, etc. | Baseline to Week 24
  Improvement of psychological statement, including sleep disorder, mood disorder, etc. is determined by the difference values of Neuropsychiatric Inventory (NPI) before and after the treatment of memantine.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided